CLINICAL TRIAL: NCT02385968
Title: Detection of Bacteria in Herniated Nucleus Material in Lumbar Disc Herniations by Culture and PCR
Status: Terminated | Type: Observational
Why Stopped: Not possible to recruit
Sponsor: Spine Centre of Southern Denmark (Other)
Collaborators: Vejle Hospital (Other)
Responsible Party: Principal Investigator, Karen Højmark Hansen, Research nurse, Sygehus Lillebaelt
Other Study IDs: S-20140085
Record Dates: First submitted 2015-03-04; First posted 2015-03-11 (Estimated); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Lumbar Disc Herniations
Keywords: Modic; Microbiology; Immunology
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsies of Nucleus
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim is to investigate if herniated nucleus material in lumbar disc herniations is infected with bacteria, and if so, to determine their prevalence (control group), and to determine if patients with pre-existing Modic changes type 1 have a higher incidence of bacterial growth in relevant lumbar disc samples than patients without Modic changes.

A cohort of 15 patients with pre-existing Modic and 15 without-undergoing primary surgery will be examined.

DETAILED DESCRIPTION:
The nucleus material will be evacuated and divided into 5 biopsies, each with a new set of sterile instruments and placed in separate sterile glass vials with one drop of sterile saline to prevent drying of biopsy.

The primary outcome, i.e., bacterial growth on a per-patient basis. Bacterial growth shall be detected in minimum 3 out of 5 biopsies for the patient to be scored as positive for bacteria.

ELIGIBILITY:
Inclusion Criteria:

* MRI-confirmed lumbar disc herniation.
* Age between 18 and 65 years.
* No prior spine surgery.
* No diagnosed dementia.

Exclusion Criteria:

* Antibiotic treatment within the previous two weeks.
* History of alcohol abuse, illicit drug use or drug abuse, or significant mental illness
* Known immune deficiency state (e.g., positive for human immunodeficiency virus) or in treatment with immunosuppressive drugs including high dose steroids or cyclosporine.
* Concurrent infections (infections of skin, urinary tract infection, other skin diseases, e.g. Acne vulgaris).
* Previous epidural instrumentation.
* Uncontrolled, unstable or recently diagnosed autoimmune disease, including but not limited to systemic lupus erythematosus, inflammatory bowel disease, sarcoidosis, rheumatoid arthritis, or psoriasis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with MRI-confirmed lumbar disc herniation. Lumbar disc herniation. Age between 18 and 65 years. No prior spine surgery. No diagnosed dementia.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Bacterial growth on a per-patient basis | at time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karen H. Hansen, Principal Investigator — Sygehus Lillebaelt
Locations (1):
- Middelfart Spinesurgery research department, Middelfart, Region Syddanmark, Denmark